CLINICAL TRIAL: NCT02238587
Title: The Effect of Gandoerma Spores Powder Capsules on the Post-treatment Life Quality and Immune Modulation of the Patients With Head-and-neck Cancer
Brief Title: The Effect of Ganoderma on Patients With Head-and-neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kuender D. Yang, MD, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 1020304
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Head-and-neck Cancer
Keywords: Gandoerma Spores Powder Capsules, head-and-neck cancer.
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/Ganoderma (Placebo Comparator): In control group, oral placebos for 6 weeks. Then the patients in control groups are switched, Ganoderma Spores Powder Capsules are given for 6 weeks. The data pertaining to their life quality are collected using Quality of Life Questionnaire after the first 6 weeks and the second 6 weeks. The immunity status is also studied at the same time.
  Interventions: Other: Control group; Dietary Supplement: Ganoderma Spores Powder Capsules
- Ganoderma (Experimental): In experimental group, Ganoderma Spores Powder Capsules for 12 weeks. The data pertaining to their life quality are collected using Quality of Life Questionnaire after the first 6 weeks and the second 6 weeks. The immunity status is also studied at the same time.
  Interventions: Dietary Supplement: Ganoderma Spores Powder Capsules

INTERVENTIONS:
Other: Control group — In control group, only placebos are given for 6 weeks. The patients who are in control groups are switched to receive Ganoderma Spores Powder Capsules for 6 weeks.
  Arms: Placebo/Ganoderma
Dietary Supplement: Ganoderma Spores Powder Capsules — In experimental group, Ganoderma Spores Powder Capsules for 12 weeks.

SUMMARY:
To study the effect of Ganoderma Spores Powder Capsules on the life quality and immunity status of the patients with head-and-neck cancer after complete treatment (including surgery and / or radiotherapy and/or chemotherapy)

DETAILED DESCRIPTION:
Ganoderma is known to modulate immunity and improve health. However, the mechanism is not clear. We hypothesize that patients who have completed standard treatment with/without radiotherapy might require biological modifier such as Ganoderma to improve life quality and immunity status.

A total of 100 patients are randomized to study and control groups. In study group, Ganoderma Spores Powder Capsules are given to the patients for 6 weeks, In control group, only placebos are given during the same period. Then the patients in study and control groups are switched, Ganoderma Spores Powder Capsules and placebos are given for 6 weeks. The data pertaining to their Life quality are collected using Quality of Life Questionnaire after the first 6 weeks and the second 6 weeks. The immunity status is also studied at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head-and-neck cancer after complete treatment for at least 3 months (including surgery and/or radiotherapy and/or chemotherapy)

Exclusion Criteria:

* Patients with head-and-neck cancer under treatment or within 3 months after treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Immune modulation such as tumor necrosis factors-α or interleukin-6 | Change from baseline in cytokines at 6 months
  Subjects will be assigned to receive placebo/Ganoderma or Ganoderma Spores Powder Capsules twice a day for 12 weeks. Peripheral blood and saliva will be collected at 3 different times: (1)baseline data: before oral intervention, (2)outcome data: at 6 and 12 weeks post-oral intervention.

SECONDARY OUTCOMES:
Life quality | Change from baseline in life quality at 6 months
  Health and life quality will assessed by Quality of Life Questionnaire at three different times: (1)baseline data: before intervention, (2)outcome data: at 6 and 12 weeks post-oral intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kuender D. Yang, PhD, Study Director — Chang Bing Show Chwan Memorial Hospital; Ching-Yeh Hsiung, Principal Investigator — Chang Bing Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan